CLINICAL TRIAL: NCT00390455
Title: Endocrine Therapy With or Without Inhibition of EGF and HER2 Growth Factor Receptors: A Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Fulvestrant With or Without Lapatinib (GW572016) for Postmenopausal Women With Hormone Receptor Positive Advanced Breast Cancer
Brief Title: Fulvestrant With or Without Lapatinib in Treating Postmenopausal Women With Stage III or Stage IV Breast Cancer That is Hormone Receptor-Positive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCI-2009-00475; NCI-2009-00475 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000510452; CALGB-40302 (Other: Alliance for Clinical Trials in Oncology); CALGB-40302 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-11

CONDITIONS: Estrogen Receptor Positive; HER2 Positive Breast Carcinoma; HER2/Neu Negative; Progesterone Receptor Positive; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Lapatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (lapatinib) (Experimental): Patients receive lapatinib ditosylate PO QD on days 1-28 and fulvestrant IM on days 1 and 15 of course 1 and on day 1 of each subsequent course. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fulvestrant; Other: Laboratory Biomarker Analysis; Drug: Lapatinib Ditosylate
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28 and fulvestrant as in Arm I. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fulvestrant; Other: Laboratory Biomarker Analysis; Other: Placebo Administration

INTERVENTIONS:
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lapatinib Ditosylate — Given PO
  Other Names: Tykerb
  Arms: Arm I (lapatinib)
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase III trial studies fulvestrant and lapatinib to see how well they work compared to fulvestrant and a placebo in treating postmenopausal women with stage III or stage IV breast cancer that is hormone receptor-positive. Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant may fight breast cancer by lowering the amount of estrogen the body makes. Lapatinib may stop the growth of breast cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether fulvestrant is more effective with or without lapatinib in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the effect, in terms of progression free survival, of the antiestrogen fulvestrant alone with fulvestrant administered in combination with the dual-kinase inhibitor lapatinib for postmenopausal women with estrogen receptor (ER) and/or progesterone receptor (PgR) positive advanced breast cancer.

SECONDARY OBJECTIVES:

I. To compare the effects of fulvestrant alone with fulvestrant and lapatinib on other clinical endpoints, including response rate, response and stable disease rate (complete response [CR] + partial response [PR] + stable disease >= 6 months), duration of response, overall survival, symptom checklist scores, and toxicity.

II. To define predictive markers of clinical activity among women receiving fulvestrant with or without lapatinib.

III. To determine if the clinical benefits for combination of hormonal and growth factor inhibitor therapy are most pronounced in women whose tumors express higher levels of ER, epidermal growth factor receptor (EGFR), human epidermal growth factor receptor 2 (HER2), phosphorylated protein kinase B (pAkt), and/or phosphorylated mitogen-activated protein kinase 1/2 (pERK1/2).

IV. To serologically determine if HER2 extracellular domain (ECD) and EGFR ECD levels can identify patients with a greater likelihood of response and clinical benefit to fulvestrant with or without lapatinib.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive lapatinib ditosylate orally (PO) once daily (QD) on days 1-28 and fulvestrant intramuscularly (IM) on days 1 and 15 of course 1 and on day 1 of each subsequent course.

ARM II: Patients receive placebo PO QD on days 1-28 and fulvestrant as in Arm I.

In both arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic, pathologic or cytologic diagnosis of cancer of the female breast in either primary or metastatic setting; histological documentation of metastatic/recurrent disease is not required if there is unequivocal clinical evidence for recurrence
* Stage IV breast cancer (using American Joint Committee on Cancer [AJCC] criteria, 6th edition), or locally advanced (stage III) breast cancer not considered amenable to curative therapy
* Patients with symptomatic brain metastases or other symptomatic central nervous system (CNS) metastases are not eligible for the study; no screening studies are required among asymptomatic patients; patients with previously treated brain metastases, who are free of symptoms referable to CNS disease and who are > 3 months from treatment for brain metastases are eligible
* Tumors (as determined on pathology from either primary or metastatic sites) must be potentially sensitive to endocrine therapy, defined as expressing estrogen receptor (ER) and/or progesterone receptor (PgR) as determined immunohistochemical methods according to the local institution's standard protocol, >= 1% cells will be considered to be positive
* The protocol has been amended to permit tumors with any HER2 status, though a determination of HER2 status must have been made; patients will be considered to be eligible if HER2 expression is documented by one of the following methods:

  * Immunohistochemistry (IHC) 0 (i.e., negative), 1+, 2+, or 3+ levels of expression, or
  * Gene amplification (fluorescent in situ hybridization [FISH]) positive or negative
* Patients must have at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2.0 cm with conventional techniques or as >= 1.0 cm with spiral computed tomography (CT) scan

  * Exception: Patients with lytic or blastic bone metastases as their only site of disease will be eligible for the study even though these patients are not considered to have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria; these patients will be evaluable for time to progression, but not response
  * Patients with all other lesions, including small lesions (longest diameter < 2.0 cm with conventional techniques or < 1.0 cm with spiral CT scan) and truly non-measurable lesions including those listed below are not eligible
  * Lesions that are considered non-measurable include the following:

    * Bone lesions (women with bone lesions will be eligible as described above)
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast cancer
    * Lymphangitis cutis/pulmonitis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Patients must have had one or two prior endocrine treatments for breast cancer in either the adjuvant or metastatic setting, exclusive of treatment-related amenorrhea or ovarian suppression; sequential use of two different third-generation aromatase inhibitors is considered "one" treatment; it is not required that tumors be resistant to such treatments; for example:

  * A patient with de novo metastatic breast cancer who had never received endocrine therapy is not eligible;
  * A patient who received adjuvant tamoxifen and subsequent therapy with an aromatase inhibitor (adjuvant or metastatic) is eligible;
  * A patient who received an aromatase inhibitor in either the adjuvant or metastatic setting, and who discontinued therapy after several months because of side effects, is eligible;
  * A patient who received an aromatase inhibitor in the adjuvant setting is eligible, regardless of whether they did or did not receive tamoxifen at some point;
  * A patient who received adjuvant tamoxifen, and subsequently a nonsteroidal aromatase inhibitor and a steroidal aromatase inhibitor for advanced breast cancer in the adjuvant or metastatic setting is eligible;
  * A patient who received adjuvant tamoxifen, and then a nonsteroidal aromatase inhibitor and subsequently megesterol acetate for advanced breast cancer is not eligible
* Tumors potentially sensitive to endocrine therapy, defined as >= 3 months of prior endocrine therapy without disease progression in the adjuvant or metastatic setting
* Patients must have had prior treatment in either the adjuvant or metastatic setting with a commercially available third-generation aromatase inhibitor (i.e. anastrozole, exemestane, or letrozole); it is not required that tumors be resistant to such therapies
* Patients may have received up to one prior chemotherapy regimen for stage IV breast cancer; prior chemotherapy in the adjuvant and/or neoadjuvant setting is permitted; patients must have finished chemotherapy at least 1 week prior to starting protocol based treatment
* Patients may have received prior trastuzumab therapy for stage IV breast cancer, in combination with up to one chemotherapy and/or endocrine therapy regimen, but that must have concluded at least 3 weeks prior to starting protocol-based therapy; prior trastuzumab therapy in the adjuvant and/or neoadjuvant setting is permitted, but must have concluded at least 3 weeks prior to starting protocol-based therapy
* Prior therapy with commercially available inhibitor of EGFR (including but not limited to gefitinib, erlotinib, lapatinib or cetuximab) or experimental inhibitors of EGFR is prohibited
* Patients may have initiated bisphosphonate therapy prior to study entry; such patients will have bone lesions considered evaluable for progression but not for response
* Prior fulvestrant therapy is prohibited
* Patients receiving a gonadotropin-releasing hormone (GnRH) agonist for ovarian suppression must remain on such therapy throughout the course of protocol treatment; patients must discontinue other endocrine treatments, including systemic hormone-replacement therapy and intravaginal estrogens prior to study entry; patients must have concluded radiation therapy prior to study entry; patients must be at least 1 week from prior chemotherapy or 3 weeks from prior trastuzumab therapy, with adequate recovery of bone marrow function and performance status
* Patients must be postmenopausal women, defined as a woman fulfilling any of the following criteria:

  * Age >= 60 years; or
  * Age >= 45 years with an intact uterus and amenorrhea for 12 months or more; or
  * History of bilateral oophorectomy; or
  * Follicle stimulating hormone (FSH) levels within postmenopausal range according to the ranges established by the testing facility; or
  * Treatment with a GnRH agonist for ovarian suppression for at least 3 consecutive months prior to study registration, and remaining on such therapy throughout the course of protocol treatment
  * Women who are pregnant or nursing are not eligible for the study; clinicians should advise patients that there are no data for the safety of lapatinib or fulvestrant among pregnant patients, nor data on the impact of these agents on fertility or pregnancy
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status 0-2
* Absence of pending visceral crisis, in the opinion of the treating physician
* Absence of acquired or inherited bleeding disorder
* Absence of need for therapeutic systemic anticoagulation (defined as maintaining international normalized ratio [INR] > 1.6); patients may take low-dose warfarin or aspirin (or equivalent) for maintenance of central venous catheter patency
* Granulocytes >= 1,000/μl
* Platelet count >= 100,000/μl
* Creatinine =< 2 mg/dl
* Total bilirubin =< 1.5 x upper limits of normal (ULN) unless due to Gilbert's syndrome
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN without liver metastases; =< 5 x ULN with liver metastases
* INR =< 1.6
* Left ventricular ejection fraction (LVEF) within institutional limits of normal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2006-09-15 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold J Burstein, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (368):
- United States (368):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arroyo Grande Community, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Saint Rose Hospital, Hayward, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Harold Leever Regional Cancer Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Portneuf Medical Center, Pocatello, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - York Hospital, York Village, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Freeman Health System, Joplin, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Saint Francis Medical Center, Trenton, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Burstein HJ, Cirrincione CT, Barry WT, Chew HK, Tolaney SM, Lake DE, Ma C, Blackwell KL, Winer EP, Hudis CA. Endocrine therapy with or without inhibition of epidermal growth factor receptor and human epidermal growth factor receptor 2: a randomized, double-blind, placebo-controlled phase III trial of fulvestrant with or without lapatinib for postmenopausal women with hormone receptor-positive advanced breast cancer-CALGB 40302 (Alliance). J Clin Oncol. 2014 Dec 10;32(35):3959-66. doi: 10.1200/JCO.2014.56.7941. Epub 2014 Oct 27. PMID 25348000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2006 and July 2010, 295 participants were recruited.
Groups:
- Arm I (Lapatinib): Patients receive 1500 mg lapatinib ditosylate PO QD on days 1-28 and fulvestrant IM on days 1 (500 mg) and 15 (250 mg) of course 1 and on day 1 (250 mg)of each subsequent course.
- Arm II (Placebo): Patients receive placebo PO QD on days 1-28 and fulvestrant IM on days 1 (500 mg) and 15 (250 mg) of course 1 and on day 1 (250 mg) of each subsequent course.
Period: Overall Study
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Started | 148 | 147
Completed | 116 | 124
Not Completed | 32 | 23
Not completed — Adverse Event | 17 | 3
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Alternate Treatment | 0 | 1
Not completed — Other Medical Reasons | 7 | 11

BASELINE CHARACTERISTICS:
Population: Four (4) participants who never started treatment were excluded from all analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo) | Total
Number analyzed (Participants) | 146 | 145 | 291
Age, Customized [Number; unit: participants]
  <40 | 8 | 7 | 15
  40-49 | 21 | 17 | 38
  50-59 | 49 | 54 | 103
  60-69 | 41 | 47 | 88
  70+ | 27 | 20 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 145 | 291
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 130 | 129 | 259
  Unknown or Not Reported | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 127 | 132 | 259
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 146 | 145 | 291
Prior tamoxifen therapy [Number; unit: participants]
  Yes | 83 | 82 | 165
  No | 63 | 63 | 126
Bond disease only [Number; unit: participants]
  Yes | 45 | 43 | 88
  No | 101 | 102 | 203

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval from study entry until disease progression or death resulting from any cause, which ever occurred first. Progression is defined as a 20% increase in the sum of longest diameter of target lesions (per RECIST criteria).
Time Frame: Interval from randomization until disease progression or death, whichever occurs first, assessed up to 5 years
Population: 4 participants who never received protocol therapy were excluded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Number analyzed (Participants) | 146 | 145
months | 4.7 [3.7 to 5.7] | 3.8 [3.8 to 5.6]
Statistical Analysis 1: Comparison: Arm I (Lapatinib) vs Arm II (Placebo); Test type: Non-Inferiority or Equivalence — The null hypothesis then is that the hazard ratio of the two treatment arms is 1.0; the alternative hypothesis is that the hazard ratio of the control to the experimental regimen is 1.5 (0.67). The test of these hypotheses is one-sided (alpha = 0.025), and interim analyses will be used to stop for futility and superiority. Under these assumptions, there is at least 90% power to detect the stated difference in median PFS between the two treatment arms; p = 0.37, Log Rank — Tests were stratified by prior tamoxifen therapy (yes/no) and bone disease only (yes/no); Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.82 to 1.33]

2. Secondary Outcome: Objective Tumor Response Rate
Description: Response was defined by the Response Evaluation Criteria in Solid Tumors (RECIST). A responding participant had either a Complete Response (disappearance of all target lesions) or Partial Response (30% decrease in sum of longest diameter of target lesions). The response rate of measurable tumors will be estimated with its 95% confidence interval according to treatment arm.
Time Frame: Up to 5 years
Population: Participants who started protocol therapy and had measurable disease were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Number analyzed (Participants) | 101 | 103
percentage of participants | 20 [13 to 29] | 9 [5 to 17]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was measured as the interval from study entry until death, from any cause, or last contact.
Time Frame: Study entry to death or last follow-up, up to 5 years
Population: 4 participants who never started protocol therapy were excluded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Number analyzed (Participants) | 146 | 145
months | 29.9 [24.8 to 34.8] | 26.4 [23.9 to 39.0]

4. Other Pre Specified Outcome: Progression-free Survival for Participants With HER2-negative Tumors
Description: PFS was defined as the interval from study entry until disease progression or death resulting from any cause, which ever occurred first.
Time Frame: Up to 5 years
Population: Participants who began protocol therapy with HER-2 negative tumors were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Number analyzed (Participants) | 122 | 113
months | 4.1 [3.4 to 5.6] | 3.8 [3.1 to 5.7]

5. Other Pre Specified Outcome: Progression-free Survival for Participants With HER2-positive Tumors
Description: PFS was defined as the interval from study entry until disease progression or death resulting from any cause, whichever occurred first.
Time Frame: Up to 5 years
Population: Participants who started protocol therapy and had HER2-positive disease were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Number analyzed (Participants) | 24 | 30
months | 5.9 [3.7 to 9.3] | 3.3 [2.1 to 7.5]

6. Other Pre Specified Outcome: Objective Tumor Response Rate for Participants With HER2-negative Tumors
Description: Response was defined by the RECIST. A responding participant had either a Complete Response (disappearance of all target lesions) or Partial Response (30% decrease in sum of longest diameter of target lesions). The response rate of measurable tumors will be estimated with its 95% confidence interval according to treatment arm.
Time Frame: Up to 5 years
Population: Participants who started protocol therapy, had measurable disease and HER-2 negative disease were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Number analyzed (Participants) | 32 | 32
percentage of participants | 13 [5 to 29] | 23 [12 to 41]

7. Other Pre Specified Outcome: Objective Tumor Response Rate for Participants With HER2-positive Tumors
Description: as for outcome 6
Time Frame: Up to 5 years
Population: Participants who started protocol therapy, had measurable disease and HER-2 positive disease were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 13
percentage of participants | 38 [14 to 70] | 17 [5 to 45]

ADVERSE EVENTS:
Description: Adverse event was available on 278 participants (Arm I: 141, Arm II: 137)
Arm/Group | Arm I (Lapatinib) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 12/141 | 14/137
Other Adverse Events (participants affected / at risk) | 128/141 | 114/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lapatinib) (N=141) | Arm II (Placebo) (N=137)
Cardiac pain (Cardiac disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 4 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (2) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (8) | 5 (5)
Gait abnormal (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 2 (2) | 3 (4)
Thrombosis (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lapatinib) (N=141) | Arm II (Placebo) (N=137)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (5) | 5 (12)
Left ventricular failure (Cardiac disorders) | 3 (6) | 3 (3)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 20 (25) | 25 (29)
Diarrhea (Gastrointestinal disorders) | 88 (206) | 30 (54)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 49 (76) | 41 (51)
Vomiting (Gastrointestinal disorders) | 22 (26) | 9 (12)
Chest pain (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 78 (205) | 73 (145)
Gait abnormal (General disorders) | 0 (0) | 1 (3)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 4 (7) | 10 (17)
Pain (General disorders) | 1 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6) | 4 (5)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (6) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (10) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 2 (2)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (4) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 19 (27) | 21 (25)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (6) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Developmental disturbance (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 19 (24) | 16 (19)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (4) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (6)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (11) | 1 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 58 (160) | 6 (16)
Rash desquamating (Skin and subcutaneous tissue disorders) | 16 (23) | 11 (13)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 38 (78) | 50 (104)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less